CLINICAL TRIAL: NCT04716283
Title: Sleep Quality and Its Determinants Among Students in Sohag University.
Brief Title: Sleep Quality Among Students in Sohag University.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Dalia Saad Louis, Demonstrator in Public Health and Community Medicine, Sohag University
Other Study IDs: soh-Med-21-01-01
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-03

CONDITIONS: Sleep

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Validated questionnaire : The Pittsburgh Sleep Quality Index (PSQI) and Epworth Sleepiness Scale (ESS) — The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score.
  The Epworth Sleepiness Scale (ESS) is a scale intended to measure daytime sleepiness .The ESS is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities.

SUMMARY:
The study will be done among undergraduate students in Sohag University for assessment of quality of sleep and its determinants .It will be done in practical faculties and theoretical faculties .

DETAILED DESCRIPTION:
Sleep is very necessary to our physical and mental health. Sleep is classified into satisfactory and unsatisfactory sleep. Good sleep is sleep which is sufficient in duration and has a good quality while bad sleep is the sleep which makes individual feels unsatisfactory .

University students are exposed to poor sleep, due to high work and study loads. Poor quality sleep has negative consequences on the daily life activities , associated with memory reduction , reduced learning abilities which ultimately can lead to reduce their academic achievements, and can also trigger negative health outcomes, such as mood disturbance, fatigue, impaired concentration .

ELIGIBILITY:
Inclusion Criteria:

* students who are in the first four years in the selected faculties .

Exclusion Criteria:

* students who will refuse to participate in this study.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will be conducted in Sohag University where there are ten practical faculties and six theoretical faculties .
  Two medical faculties and two non medical faculties were chosen randomly to be the setting of the study.
Sampling Method: Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-08-26 (Estimated); Study Completion 2022-10-10 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index [PSQI] | It will be measured after completion of the study ,approximately in october 2022.
  A questionnaire will be used to measure sleep quality over the last 1 month .The self-related questions include the assessment of seven different sleep domains : sleep quality, sleep latency , sleep duration , habitual sleep efficiency, sleep disturbances , use of sleeping medications , and daytime dysfunction .The seven components scores are then added to yield a global PSQI score in the range of zero to 21. The higher the score, the worse the sleep quality. A global score greater than five is diagnostic of poor sleep quality.
Epworth Sleepiness Scale [ESS] | It will be measured after completion of the study ,approximately in octuber 2022.
  A questionnaire will be used to measure daytime sleepiness .It can determine the chance of falling asleep in 8 different circumstances. ESS score can range from 0 to 24. A global score greater than ten is diagnostic of excessive daytime sleepiness .

CONTACTS AND LOCATIONS:
Overall Officials: Dalia S Louis, Demonstrator, Principal Investigator — Faculty of Medicine -Sohag University
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No